CLINICAL TRIAL: NCT06657417
Title: A.I. Supported Laryngoscopy and Endotracheal Intubation: a Manikin Study
Acronym: aiTN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Schulthess Klinik (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ANEST-0004
Record Dates: First submitted 2024-09-03; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Intubation; Difficult or Failed
Keywords: Tracheal intubation; airway management; C-MAC video laryngoscope; LarynGuide software

STUDY DESIGN:
Intervention Model Description: The trial is a randomized 2x2 crossover design. Each procedure will be performed by the same participant in sequence with at least 3 days between the first and second round of procedures. The procedures will be performed in sequence to which the participants were randomized (TC: First Test and then Control or CT: First Control and then Test). A sequence of 6 intubations will be performed in each sitting (in order, 3 easy and 3 difficult).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard before AI support (Experimental)
  Interventions: Device: Video laryngoscopy
- AI support before standard (Experimental)
  Interventions: Device: Video larnygoscopy

INTERVENTIONS:
Device: Video laryngoscopy — Standard video laryngoscopy before video laryngoscopy with additional larynGuide overlay
  Arms: Standard before AI support
Device: Video larnygoscopy — Video laryngoscopy with additional larynGuide overlay before standard video laryngoscopy
  Arms: AI support before standard

SUMMARY:
LarynGuide is a newly developed AI-supported software for video laryngoscopy that supports the user through correct placement of endotracheal tube by means of audio-visual signals and warning of incorrect or potentially dangerous handling. This prospective study assesses the performance of tracheal intubation using video laryngoscopy with larynGuide AI overlay as compared to standard video larnygoscopy an simulation setting.

DETAILED DESCRIPTION:
Tracheal intubation is a core competence in anesthesia and emergency medicine. This complex medical procedure aims to preserve gas exchange in the lungs. Vital for that is a secured and patent airway as soon as spontaneous ventilation ceases under general anesthesia or in life-threatening conditions like (e.g, respiratory insufficiency or resuscitation). Failure in securing an airway can result in hypoxemia, leading to neurologic damage, cardiovascular complications, and death. Complex anatomic structures or abnormalities of the upper airway, as well as airway trauma, bear the risk of failed intubation and inability to ventilate the lungs, which furthermore may result in ventilation and oxygenation failure. Tracheal intubation's success highly depends on user experience and skills. Literature reports unexpected difficult intubations ranging from 5 to 10%, mostly corresponding to a Cormack/Lehane grade 3 or 4.4-7. Besides classic direct laryngoscopes and flexible optic endoscopes, video laryngoscopes with high-resolution video cameras placed at the tip of the devices facilitate tracheal intubation. Video laryngoscopy seems superior in normal and difficult intubation, as it improves the first-attempt success rate.

Complication rates and upper airway trauma after direct laryngoscopy with a Macintosh type blade in patients with normal airway have been reported up to 7%15. Video laryngoscopy reduces that relative high incidence Upper airway trauma is increased when physical force is used during laryngoscopy to improve limited view on the glottis16 or if more than two intubation attempts are needed. The newly developed larynGuide software is an artificially intelligent video laryngoscope monitoring system which provides information to the user on visible anatomy, next steps to advance the oro-tracheal intubation to completion, and to advise on un-safe or incorrect maneuvers & interventions. As soon as the device places the scope into the trachea the provider slides the tracheal tube over the scope into the proper place of the trachea as usually done during flexible scope intubation.

Aimof this study is to determine the effects larynGuide has on tracheal intubation performance compared with standard of care video laryngoscopy.

ELIGIBILITY:
1. Volunteer medical professionals
2. Experienced: consultant anaesthetists, resident anaesthetists and certified nurse
3. Inexperienced: junior doctors (other than anaesthetists), clinical year medical students, nurses and paramedics

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-08-25 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Rate of first-attempt tracheal intubation success | 2 minutes
  12 single attempts per participant

SECONDARY OUTCOMES:
Time to intubation | 2 minutes
  12 single attempts per participant
Rate of total intubation success | 2 minutes
  12 single attempts per participant
Global Rating Scale of Procedural Performance | 2 minutes
  instrument handling, flow and knowledge of procedure for each intubation on a grade scale from 1 to 5; 12 single time points per participant
Percentage of dental damage incidence | 2 minutes
  12 single attempts per participant

CONTACTS AND LOCATIONS:
Overall Officials: Christoph K Hofer, MD, Study Chair — Schulthess Klinik
Locations (1):
- Schulthess Klinik, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No